CLINICAL TRIAL: NCT02025335
Title: Assessment of CMV-specific ELISPOT Assay for Predicting CMV Infection in Kidney Transplant Recipients (ACE-KT)
Brief Title: Assessment of CMV-specific ELISPOT Assay for Predicting CMV Infection in Kidney Transplant Recipients
Acronym: ACE-KT
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sung-Han Kim, Associate Professor, Asan Medical Center
Other Study IDs: 2013-1040; 2013-1040
Record Dates: First submitted 2013-12-16; First posted 2014-01-01 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Kidney Transplantation Recipients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- high CMV ELISPOT results: high spot counts in ELISPOT
- low CMV ELISPOT results: low spot counts in ELISPOT

SUMMARY:
CMV is one of the most important opportunistic infection in transplant recipients. In South Korea, more than 95% of adults reveal sero-positivity for CMV IgG. Until now, sero-positivity for CMV IgG before solid organ transplantation is a laboratory test of choice to stratify the risk of CMV reactivation after solid organ transplantation. Theoretically, CMV-specific cell-mediate immune response before solid organ transplantation will further categorize the patients into high or low risk of CMV development after solid organ transplantation. The investigators thus evaluate the usefulness of CMV-specific ELISPOT assay in kidney transplant candidates to predict the development of CMV infection after kidney transplantation.

DETAILED DESCRIPTION:
Between Mar 2014 and Mar 2015, all patients admitted in the kidney transplant unit will be enrolled in this study. All patients will receive CMV-specific ELISPOT assay and be prospectively followed for the development of CMV infection.

ELIGIBILITY:
Inclusion Criteria:

* age 16 or more
* agree with written informed consent

Exclusion Criteria:

* donor CMV IgG (+) and recipient CMV IgG (-)

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kindeny transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
CMV infection | 6 months after transplantation
  CMV infection is defined as follows.
  1. CMV viremia: CMV antigenemia or CMV quantitative PCR (+)
  2. CMV disease: CMV syndrome or tissue-invasive CMV disease i) CMV syndrome: ① CMV viremia ② temperature > 38 without other cause ③ WBC < 4000, atypical lymphocyte > 3%, transaminase elevation, platelet < 100,000/mm ii) tissue-invasive CMV disease: evidence of CMV in histopathologic specimen (inclusion body or viral antigen in biopsy or bronchoalveolar lavage fluid)

SECONDARY OUTCOMES:
mortality | 6 months after transplantation
rejection | 6 months after transplantation
graft loss | 6 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Han Kim, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim T, Lee HJ, Kim SM, Jung JH, Shin S, Kim YH, Sung H, Chong YP, Lee SO, Choi SH, Kim YS, Woo JH, Kim SH, Han DJ. Diagnostic usefulness of the cytomegalovirus (CMV)-specific T cell-based assay for predicting CMV infection after kidney transplant. Korean J Intern Med. 2020 Mar;35(2):438-448. doi: 10.3904/kjim.2017.318. Epub 2018 Jun 7. PMID 29865778